CLINICAL TRIAL: NCT03430622
Title: Telephone Delivered Learning Through Play (LTP) Plus Interpersonal Psychotherapy (IPT) for Depressed Mothers - A Multicentre Randomized Controlled Trial (RCT) in a Low-Income Country
Brief Title: Learning Through Play (LTP) Plus Interpersonal Psychotherapy (IPT)
Acronym: TLMC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pakistan Institute of Living and Learning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PILL-Telemothercare01
Record Dates: First submitted 2018-02-06; First posted 2018-02-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Maternal Depression
MeSH Terms: interventions — Long-Term Potentiation; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Researchers doing outcome assessment will be kept blind to the group allocations
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTP Plus (Experimental): LTP Plus group participants will receive intervention over the telephone for 3 months one session per week for 2 months and rest of the sessions fortnightly by trained graduates, expert in delivering LTP plus intervention.
  Interventions: Behavioral: LTP Plus
- Treatment as Usual (TAU) (Active Comparator): TAU group will receive routine care and their follow up will be done after completion of the intervention and then at 6-month post randomization.
  Interventions: Other: TAU

INTERVENTIONS:
Behavioral: LTP Plus — LTP Plus is comprised of two components; Learning through play (LTP) and Interpersonal Psychotherapy (IPT). The LTP Plus is a low-literacy; sustainable program intended to provide parents with information on the healthy growth and development of their young children. The LTP research-based activities enhance children's development while simultaneously promoting attachment security through building parents' ability to read and be sensitive to their children's cues and through active involvement in their children's development. Plus the Interpersonal Psychotherapy (IPT) intervention is comprised of a supportive element, an educational element, a parenting element and an interpersonal relationship element. Intervention goals include helping mothers feel supported, empowered and confident about their parenting abilities, which would directly influence reduction in depressive symptoms as well as resolution of interpersonal conflicts.
  Other Names: Psycho-social Intervention
  Arms: LTP Plus
Other: TAU — This group will be on their routine care and will not be given any intervention
  Other Names: Treatment as Usual
  Arms: Treatment as Usual (TAU)

SUMMARY:
To evaluate the effectiveness of a telephone based LTP Plus intervention for maternal depression.

DETAILED DESCRIPTION:
Despite the high prevalence of maternal depression in Pakistan, research on psychosocial interventions is limited. We will test the effectiveness of a telephone based intervention program called Learning through Play plus Interpersonal Psychotherapy (LTP Plus) that can be used by non-specialists, including trained graduates, mothers and lay health workers with minimal training. This telephone communication will be supplemented by the provision of LTP Plus pictorial calendars to the depressed mothers.

Purpose of this RCT is to determine if telephone delivered intervention of the LTP plus programme reduces symptoms of maternal depression and improves infant development compared to Treatment as usual. A sample of 354 (177 in each group) will be required. The study will be conducted in big cities of Pakistan including Karachi, Lahore, Hyderabad, Nawabshah, Quetta and Peshawar.Participants will be screened using Patient Health Questionnaire (PHQ-9) and eligibility checklist. Those scoring 10 and above on PHQ-9 will be invited to participate in the study. Assessments will be done at baseline and after completion of intervention (3rd month and 6th month after randomization). All follow ups will be done by independent Research Assistants (RAs), blind to the treatment allocations.

ELIGIBILITY:
Inclusion Criteria:

Participants will be included in the study if they are:

18 to 44 years old mothers with children aged between 0-30 months having a diagnosis of major depressive disorder using the Structure Clinical Interview for DSM-V, Ability to complete a baseline assessment, Participating mother having telephone/mobile phone access for at least one hour per week.

Exclusion Criteria:

Participants will be excluded from the study if they have:

Any medical illness that will prevent them from participation in the clinical trial, current or past diagnosis of bipolar depression, currently using antidepressants or receiving any kind of psychotherapy, active suicidal ideation, any other severe physical or mental disorder, no access to telephone/mobile.

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 370 (Actual)
Dates: Start 2018-02-20 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Structured Clinical Interview for DSM-IV (SCID) | Time Frame: Changes from baseline to 6th month after randomization ]
  The primary outcome is depression which will be measured using Structured Clinical Interview for DSM-V Disorders (SCID)

SECONDARY OUTCOMES:
Generalized Anxiety Disorder (GAD) 7 | [Time Frame: Changes from baseline to 3rd month and 6th month after randomization]
  The GAD-7 is a 7 item scale will be used to screen for and measure severity of Generalized Anxiety Disorder
The Postpartum Bonding Questionnaire (PBQ) | [Time Frame: Changes from baseline to 3rd month and 6th month after randomization]
  The PBQ is designed to detect disturbance in the mother-child relationship. The scale has 25 items, each followed by six alternative responses ranging from 'always' to 'never'.
Experiences in Close Relationships-Revised (ECR-R) | [Time Frame: Changes from baseline to 3rd month and 6th month after randomization]
  The ECR-R measures individuals on two subscales of attachment: Avoidance and Anxiety. In general avoidant individuals find discomfort with intimacy and seek independence, whereas anxious individuals tend to fear rejection and abandonment.
Dyadic Adjustment Scale, (DAS) | [Time Frame: Changes from baseline to 3rd month and 6th month after randomization]
  DAS is a 32 items self-report questionnaire, to measure couple satisfaction and to assess how each partner perceives his/her relationship.
Client Service Receipt Inventory | [Time Frame: Changes from baseline to 3rd month]
  We will collect information about the use of other health services (including the informal sector, faith healers/Imams) using CSRI based on our previous work in Pakistan.
Infant development: Infant development: | [Time Frame: Changes from baseline to 3rd month and 6th month after randomization]
  Ages and Stages Questionnaire will be used to measure child development. Parents will report on their child's communication, gross and fine motor skills, problem solving and personal-social development at different time points.
Ages and Stages Social-Emotional Questionnaire | Changes from baseline to 3rd month and 6th month after randomization]
  Ages and Stages will be used to obtain maternal report on their child's social and emotional development. The questionnaire is already translated in Urdu and will be used in the proposed trial.
World Health Organisation Quality of Life (WHO, 2004) | Changes from baseline to 3rd month and 6th month after randomization]
  A self-report scale comprising of 26 items which measures physical health, psychological health, social relationships and environment.
Learning Through Play (LTP) KAP Questionnaire | Changes from baseline to 3rd month and 6th month after randomization]
  This scale will be used to measure change in Knowledge, Attitude and Practices (KAP) at different time points.
Patient Health Questionnaire (PHQ-9) | Time Frame: Changes from baseline to 3rd month and 6th month after randomization ]
  The Patient health Questionnaire (PHQ-9) is 9 items self-report questionnaire. A score of 10 or above is taken as cut -off point for depressive disorder. This scale will be used to check severity of depression.
  Patient Health Questionnaire (PHQ-9) The Patient health Questionnaire (PHQ-9) is 9 items self-report questionnaire. A score of 10 or above is taken as cut -off point for depressive disorder. This scale will be used to check severity of depression.
Client Satisfaction Questionnaire | Time Frame: Score at 3rd month assessment only.
  The participants will rate their satisfaction with treatment after completion of intervention. Higher score indicate greater satisfaction
How are you feeling scale | Time Frame: Changes from baseline to 3rd month and 6th month after randomization ]
  This is a pictorial scale to assess mood disturbance. higher score indicate greater severity of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nasim Chaudhry, Principal Investigator — Pakistan Institute of Living & Learning
Locations (6):
- Pakistan (6):
  - Pediatric units, Quetta, Balochistan
  - Pedratric units, Lahore, Punjab Province
  - Pediatric units, Hyderābād, Sindh
  - Pediatric units, Karachi, Sindh
  - Pediatric units, Nawabshah, Sindh
  - Pediatric units, Peshawar, Sindh

IPD SHARING:
Plan to Share IPD: No